CLINICAL TRIAL: NCT05394961
Title: Are Socioeconomic Factors, Sex and Country of Birth Associated With Decisions to Withhold or Withdraw Intensive Care in Swedish Hospitals?
Brief Title: Factors Associated With Decisions to Withhold or Withdraw Intensive Care
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: Uppsala University
Record Dates: First submitted 2022-05-23; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Sepsis; ARDS, Human; COVID-19
Keywords: critical care; limitations of care; critical illness; intensive care unit
MeSH Terms: conditions — Sepsis; Respiratory Distress Syndrome; COVID-19; Critical Illness | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Treatment in an intensive care unit with a diagnosis of sepsis and/or ARDS and/or covid-19 — As above

SUMMARY:
Medical and socioeconomic data are extracted from the Swedish Intensive Care Registry (SIR), the Swedish National Patient Registry and Statistics Sweden for all adult patients admitted to in Swedish intensive care units between 2014-01-01 and 2020-12-31 with a diagnosis of sepsis and/or acute respiratory distress syndrome (ARDS) and/or coronavirus 19 (COVID-19) infection, and registered in SIR. The impact of demographic and socioeconomic factors on decisions to withhold or withdraw intensive care, and on mortality, are studied and statistically adjusted for level of chronic comorbidity and severity of acute illness.

DETAILED DESCRIPTION:
Patient identification and data acquisition With permission from the ethical board of Sweden, all registered intensive care episodes with a diagnosis of sepsis, acute respiratory distress syndrome (ARDS) or coronavirus 19 (COVID-19) and admission between 2014-01-01 and 2020-12-31 are identified in the Swedish Intensive Care Registry (SIR). Basic demographic data (age, sex) and intensive care data from SIR are combined with comorbidity data from the National Patient Registry of the Board of Health and Welfare (Socialstyrelsen), and data on country of birth, household size, education and economy from Statistics Sweden (SCB) to produce a pseudonymized study data set. For patients with multiple intensive care episodes, the first one is used.

Analysis Descriptive data on the frequency of decisions to withhold or withdraw intensive care, and on demographic and socioeconomic factors, morbidity and mortality in patients with or without such decisions, are produced. Logistic regression is used to assess the association between demographic and socioeconomic factors and limitations in intensive care, adjusting for acute and chronic morbidity and accounting for multicenter data. Secondarily, association between the same factors and mortality is studied.

ELIGIBILITY:
Inclusion Criteria:

* Registered intensive care episode with relevant diagnosis

Exclusion Criteria:

* None, if inclusion criteria fulfilled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of an absolute majority of the patients treated in Swedish intensive care units with the relevant diagnoses during the study period and can therefore be considered a nationwide population rather than a sample thereof.
Sampling Method: Non-Probability Sample
Enrollment: 33256 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Decision to withhold or withdraw intensive care | During ICU care
  Registered decision

SECONDARY OUTCOMES:
30 day mortality | 30 days
  death within 30 days of ICU admission
90 day mortality | 90 days
  death within 90 days of ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Miklós Lipcsey, MD, PhD, Principal Investigator — Upsala University
Locations (1):
- Uppsala University, department of Surgical Sciences, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data are used with special permission from the national ethical bord of Sweden (Etikprövningsmyndigheten) and the involved register keepers and so cannot be shared without an extended permission.